CLINICAL TRIAL: NCT03741881
Title: A Prospective, Multi-national, Non-interventional Study in Haemophilia A and B Patients With or Without Inhibitors Treated According to Routine Clinical Treatment Practice (Explorer™6)
Brief Title: A Study Following People With Haemophilia A and B, With or Without Inhibitors, When on Usual Treatment (Explorer™6)
Acronym: explorer™6
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7415-4322; U1111-1182-3359 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Haemophilia A; Haemophilia A With Inhibitors; Haemophilia B; Haemophilia B With Inhibitors
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haemophilia: Patients with haemophilia A or B and with or without inhibitors
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Participants are treated with their usual prescribed treatment, either given regularly as a prevention (prophylaxis) or when needed (on-demand).

SUMMARY:
This study will collect data on bleeds and data related to quality of life in people with severe congenital (a disease existing from birth) haemophilia A and B, with or without inhibitors. The aim for the study is to look at the number of bleeds when on usual treatment for haemophilia. Participants will be asked to keep an electronic diary to track the number of bleeds and the treatment of their bleeds. Participants will be asked to wear an activity tracker on their wrist to capture their level of activity every day for up to 12 weeks. While taking part in this study, participants will keep getting their usual treatment as given to them by their doctor. All study visits at the clinic are done in the same way as the participants are used to. In the time between the participants' visits to the clinic, the study staff at the clinic may call or email the participant. The study will last for about 2½ years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine eligibility for the study.
2. Male, age equal to or above 12 years at the time of signing informed consent.
3. Patients with congenital haemophilia with inhibitors treated with FEIBA® prophylaxis: equal to or above 2 treated bleeding episodes within 24 weeks before screening (visit 1).

   (For Turkey only: Patients with congenital haemophilia with inhibitors treated with by-passing agents prophylaxis: equal to or above 2 treated bleeding episodes within 24 weeks before screening (visit 1)).
4. Severe (FVIII activity below 1%) congenital haemophilia A or severe/moderate (FIX activity equal to or below 2%) congenital haemophilia B, or congenital haemophilia A or B of any severity, with a presence or history of inhibitor (equal to or above 0.6 Bethesda Unit (BU)), based on medical records
5. Patients with CHwI treated on-demand: equal to or above 6 treated (with bypassing agent) bleeding episodes within 24 weeks (or equal to or above 12 during 52 weeks) before screening (visit 1) and patients with severe congenital HA/HB treated on-demand: equal to or above 5 treated (with factor product) bleeding episodes within 24 weeks (or equal to or above 10 during 52 weeks) before screening (visit 1).

Exclusion Criteria:

1. Known or suspected hypersensitivity to monoclonal antibodies.
2. Previous participation in this study. Participation is defined as signed informed consent.
3. Any disorder, except for conditions associated with congenital haemophilia, which in the physician's opinion might jeopardise patient's safety or compliance with the protocol.
4. Previous treatment with concizumab. Previous treatment is defined as two or more doses administered.
5. Planned FVIII/FIX Immune Tolerance Induction (ITI) regimens during the study.
6. Current or planned treatment with emicizumab.
7. Any known congenital or acquired coagulation disorder other than congenital haemophilia.
8. History of thromboembolic disease, current clinical signs of or treatment for thromboembolic disease, or at high risk of thromboembolic disease as judged by the investigator.
9. Presence or history of malignant neoplasm within 5 years prior to the day of screening.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia A or B and with or without inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
The number of treated bleeding episodes | From enrolment (week 0) and up to a maximum of 115 weeks
  Count of treated bleeding episodes

SECONDARY OUTCOMES:
The number of all bleeding episodes | From enrolment (week 0) and up to a maximum of 115 weeks
  Count of bleeding episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (129):
- United States (27):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Macon, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, East Lansing, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Algeria (2):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Constantine
- Australia (3):
  - Novo Nordisk Investigational Site, Melbourne, Victoria
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Murdoch, Western Australia
- Novo Nordisk Investigational Site, Amstetten, Austria
- Novo Nordisk Investigational Site, Banja Luka, Bosnia and Herzegovina
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Canada (4):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Saint John, New Brunswick
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Hamilton, Ontario
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Tallinn, Estonia
- Novo Nordisk Investigational Site, Helsinki, Finland
- France (9):
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Saint-Etienne
- Germany (2):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Homburg
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Novo Nordisk Investigational Site, Budapest, Hungary
- India (5):
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (5):
  - Novo Nordisk Investigational Site, Castelfranco Veneto
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Udine
  - Novo Nordisk Investigational Site, Verona
- Japan (13):
  - Novo Nordisk Investigational Site, Aichi
  - Novo Nordisk Investigational Site, Hiroshima
  - Novo Nordisk Investigational Site, Hyōgo
  - Novo Nordisk Investigational Site, Kagoshima
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kyoto
  - Novo Nordisk Investigational Site, Mie
  - Novo Nordisk Investigational Site, Nara
  - Novo Nordisk Investigational Site, Niigata
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Saitama
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Novo Nordisk Investigational Site, Selangor Darul Ehsan, Malaysia
- Novo Nordisk Investigational Site, Monterrey, Nuevo León, Mexico
- Novo Nordisk Investigational Site, Groningen, Netherlands
- Novo Nordisk Investigational Site, Oslo, Norway
- Poland (3):
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Warsaw
- Novo Nordisk Investigational Site, Porto, Portugal
- Russia (3):
  - Novo Nordisk Investigational Site, Krasnodar
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Novi Sad
- Novo Nordisk Investigational Site, Bratislava, Slovakia
- South Africa (3):
  - Novo Nordisk Investigational Site, Parktown, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Polokwane, Limpopo
- South Korea (4):
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Daejeon
  - Novo Nordisk Investigational Site, Jeju-do
  - Novo Nordisk Investigational Site, Seoul
- Spain (5):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Oviedo
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Sweden (2):
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Solna
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Turkey (Türkiye) (8):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Capa-ISTANBUL
  - Novo Nordisk Investigational Site, Edirne
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Samsun
- Ukraine (2):
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Lviv
- United Kingdom (6):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Wheeler AP, Abraham A, Barnes C, Brown Frandsen R, d'Oiron R, Eichler H, Hampton K, Lopez-Jaime FJ, Lyu CJ, Tavares CMM, Nogami K, Sutton C, Windyga J, Zulfikar B, Castaman G. Real-World Unmet Needs of Patients With Haemophilia A and Haemophilia B With or Without Inhibitors: End-of-Study Results From the explorer6 Non-Interventional Study. Haemophilia. 2025 Sep;31(5):903-911. doi: 10.1111/hae.70051. Epub 2025 May 5. PMID 40323006